CLINICAL TRIAL: NCT03254290
Title: Color Stability of NeoMTA Pulpotomized Primary Teeth
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas A & M University Baylor College Of Dentistry (Other)
Responsible Party: Principal Investigator, Carolyn A. Kerins DDS, Principal Investigator, Texas A & M University Baylor College Of Dentistry
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TexasAMBaylor
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Dental Caries Extending to Pulp
MeSH Terms: interventions — formocresol

STUDY DESIGN:
Intervention Model Description: Children between the ages of 2 ½ and 9 years of age and be ASA I or ASA II. Patient must have two, primary teeth that are matched for, size of carious lesion (same level of approximation of carious lesion to the pulp) and are that are treatment planned for a pulpotomy. The teeth selected for the study must be vital and asymptomatic both clinically and radiographically or only display symptoms consistent with reversible pulptitis The teeth selected for the study must be anticipated to be retained in the mouth for at least eighteen months
Who Masked: Participant
Masking Description: The teeth treated with each specific material will be randomly assigned by drawing a random number from a manilla folder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental NeoMTA (Experimental): The new formulation of MTA (does not contain bismuth oxide) will be used in one tooth receiving a pulpotomy to determine if the color of the tooth changes over time.The new formulation has received the FDAs 510(k) substantial equivalence clearance for Class II dental materials and is equivalent to its MTA predicate (ProRoot, Dentsply Tulsa Dental, Tulsa, OK, USA).
  Interventions: Biological: NeoMTA; Biological: Formocresol
- Formocresol (Active Comparator): Control group. This group will receive the "gold standard" formulation of a formocresol pulpotomy.
  Interventions: Biological: Formocresol

INTERVENTIONS:
Biological: NeoMTA — A new formulation of MTA was developed in which bismuth oxide was omitted.
  Arms: Experimental NeoMTA
Biological: Formocresol — Control group

SUMMARY:
This randomized control study will use 15 pediatric subjects selected from the patient population in the pediatric dental clinic at Children's Medical Center Dental Clinic (CMC Dental Clinic). The study will use a within-subject control design whereby one tooth will be treated with a pulpotomy using the new formulation of MTA (NeoMTA Plus, Avalon Biomed Inc., Bradenton, FL, USA) and restored with a multi-surface composite, and the other tooth with a formocresol pulpotomy and restored with a multi-surface composite; thus, approximately 15 teeth will be treated for each treatment group. The specific treated tooth will be randomized as to which side will receive the MTA or formocresol using sealed, opaque envelopes. Approximately 15 subjects will be needed for the study in order to elicit any significant findings as demonstrated by a power analysis.

DETAILED DESCRIPTION:
Each of the 15 patients will represent a pair of teeth. Within a given patient, assignment of the first tooth to either treatment will be determined randomly by selecting a sealed, opaque envelope with a designated treatment, with another tooth being assigned to the other treatment. All patients must demonstrate sufficient cooperation for treatment and follow-up radiographs. All procedures, possible risks or discomforts, in addition to possible benefits will be explained to the parents of all patients involved, and informed consent will be obtained from each parent.

The goal will consist of completing all treatment in one appointment; however, in the event that all treatment is unable to be completed, for example, local anesthetic limitations, the patient will be scheduled for the next available appointment, keeping them as close together as possible.

Patients will be anesthetized with local anesthesia, and treatment will be performed utilizing rubber dam isolation. The pulpotomy procedure will include removal of the carious tooth structure using a high-speed carbide bur and water spray. When the removal of carious tooth structure results in pulp exposure, the roof of the chamber will be removed. A high-speed handpiece and sterile spoon excavator will be used to remove the coronal pulp tissue. The amputation site will be cleaned and hemostasis obtained with a wet cotton pellet. The site will then be treated with either a slurry of NeoMTA Plus according to the manufacturer's directions or traditional Formocresol according to the manufacturer's directions. The remaining pulp chamber will be filled with a visible light cured resin-reinforced glass ionomer and will then receive a multi-surface composite final restoration

ELIGIBILITY:
Inclusion Criteria:

Children between the ages of 2 ½ and 9 years of age and be ASA I or ASA II. Patient must have two, primary teeth that are matched for, size of carious lesion (same level of approximation of carious lesion to the pulp) and are that are treatment planned for a pulpotomy. The teeth selected for the study must be vital and asymptomatic both clinically and radiographically or only display symptoms consistent with reversible pulptitis The teeth selected for the study must be anticipated to be retained in the mouth for at least eighteen months

Exclusion Criteria:

Teeth with a history of spontaneous pain. Teeth with radiographic evidence of internal or external resorption, intraradicular or periapical bone loss, loss of lamina dura, or widening of the periodontal ligament space

Ages: 30 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Color stability | 3 month recall
  color scale (0=white/still esthetic; 1=slightly gray; 2=medium gray color; 3=dark gray

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Agamy HA, Bakry NS, Mounir MM, Avery DR. Comparison of mineral trioxide aggregate and formocresol as pulp-capping agents in pulpotomized primary teeth. Pediatr Dent. 2004 Jul-Aug;26(4):302-9. PMID 15344622
- [Result] Farsi N, Alamoudi N, Balto K, Mushayt A. Success of mineral trioxide aggregate in pulpotomized primary molars. J Clin Pediatr Dent. 2005 Summer;29(4):307-11. doi: 10.17796/jcpd.29.4.n80t77w625118k73. PMID 16161395
- [Result] Holan G, Eidelman E, Fuks AB. Long-term evaluation of pulpotomy in primary molars using mineral trioxide aggregate or formocresol. Pediatr Dent. 2005 Mar-Apr;27(2):129-36. PMID 15926290
- [Result] Jabbarifar SE, Khademi D, Ghasemi D. Success rates of formocresol pulpotomy versus mineral trioxide aggregate in human primary molar tooth. J Res Med Sci 2004; 9(6)L 55-8.
- [Result] Peng L, Ye L, Tan H, Zhou X. Evaluation of the formocresol versus mineral trioxide aggregate primary molar pulpotomy: a meta-analysis. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Dec;102(6):e40-4. doi: 10.1016/j.tripleo.2006.05.017. Epub 2006 Sep 26. PMID 17138165
- [Result] Farooq NS, Coll JA, Kuwabara A, Shelton P. Success rates of formocresol pulpotomy and indirect pulp therapy in the treatment of deep dentinal caries in primary teeth. Pediatr Dent. 2000 Jul-Aug;22(4):278-86. PMID 10969431
- [Result] Guelmann M, Fair J, Bimstein E. Permanent versus temporary restorations after emergency pulpotomies in primary molars. Pediatr Dent. 2005 Nov-Dec;27(6):478-81. PMID 16532888
- [Result] Holan G, Fuks AB, Ketlz N. Success rate of formocresol pulpotomy in primary molars restored with stainless steel crown vs amalga. Pediatr Dent. 2002 May-Jun;24(3):212-6. PMID 12064493
- [Result] Seale NS. The use of stainless steel crowns. Pediatr Dent. 2002 Sep-Oct;24(5):501-5. PMID 12412965
- [Result] Caceda JH. The use of resin-based composite restorations in pulpotomized primary molars. J Dent Child (Chic). 2007 May-Aug;74(2):147-50. PMID 18477438
- [Result] Cehreli ZC, Cetinguc A, Cengiz SB, Altay AN. Clinical performance of pulpotomized primary molars restored with resin-based materials. 24-month results. Am J Dent. 2006 Oct;19(5):262-6. PMID 17073200
- [Result] Guelmann M, Bookmyer KL, Villalta P, Garcia-Godoy F. Microleakage of restorative techniques for pulpotomized primary molars. J Dent Child (Chic). 2004 Sep-Dec;71(3):209-11. PMID 15871455
- [Result] Guelmann M, McIlwain MF, Primosch RE. Radiographic assessment of primary molar pulpotomies restored with resin-based materials. Pediatr Dent. 2005 Jan-Feb;27(1):24-7. PMID 15839391
- [Result] Hutcheson C, Seale NS, McWhorter A, Kerins C, Wright J. Multi-surface composite vs stainless steel crown restorations after mineral trioxide aggregate pulpotomy: a randomized controlled trial. Pediatr Dent. 2012 Nov-Dec;34(7):460-7. PMID 23265162
- [Result] Maroto M, Barberia E, Planells P, Garcia Godoy F. Dentin bridge formation after mineral trioxide aggregate (MTA) pulpotomies in primary teeth. Am J Dent. 2005 Jun;18(3):151-4. PMID 16158803
- [Result] Parirokh M, Asgary S, Eghbal MJ, Stowe S, Eslami B, Eskandarizade A, Shabahang S. A comparative study of white and grey mineral trioxide aggregate as pulp capping agents in dog's teeth. Dent Traumatol. 2005 Jun;21(3):150-4. doi: 10.1111/j.1600-9657.2005.00311.x. PMID 15876326
- [Result] Holland R, de Souza V, Murata SS, Nery MJ, Bernabe PF, Otoboni Filho JA, Dezan Junior E. Healing process of dog dental pulp after pulpotomy and pulp covering with mineral trioxide aggregate or Portland cement. Braz Dent J. 2001;12(2):109-13. PMID 11445912
- [Result] Maroto M, Barberia E, Vera V, Garcia-Godoy F. Dentin bridge formation after white mineral trioxide aggregate (white MTA) pulpotomies in primary molars. Am J Dent. 2006 Apr;19(2):75-9. PMID 16764128
- [Result] Walsh RM, Woodmansey KF, Glickman GN, He J. Evaluation of compressive strength of hydraulic silicate-based root-end filling materials. J Endod. 2014 Jul;40(7):969-72. doi: 10.1016/j.joen.2013.11.018. Epub 2014 Jan 14. PMID 24935545
- See also: Avalon Biomed Inc 2014 — http://www.accessdata.fda.gov/cdrh_docs/pdf14/K140955.pdf